CLINICAL TRIAL: NCT03560947
Title: Modelo Preditivo Para os Resultados de Sucesso Com um Programa Combinado de Terapia Manual e exercício em indivíduos Com Dor Cervical crónica de Origem não-especifica
Brief Title: Individual Responder Analysis of the Effectiveness of Manual Therapy and Exercise Versus Usual Care in Patients With Chronic Nonspecific Neck Pain
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Universidade Nova de Lisboa (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: NMS|FCM-UNL
Record Dates: First submitted 2018-05-23; First posted 2018-06-18 (Actual); Last update posted 2018-06-18 (Actual); Status verified 2018-06

CONDITIONS: Chronic Nonspecific Neck Pain
Keywords: chronic nonspecific neck pain; exercise; manual therapy
MeSH Terms: conditions — Motor Activity | interventions — Musculoskeletal Manipulations; Exercise

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Manual Therapy and Exercise (Experimental)
  Interventions: Other: Manual Therapy and Exercise (Physiotherapy Intervention)
- Usual Care (Active Comparator)
  Interventions: Other: Usual Care (Physiotherapy Intervention)

INTERVENTIONS:
Other: Manual Therapy and Exercise (Physiotherapy Intervention) — Experimental group: Manual Therapy and Exercise Participants in this group will receive a 6-weeks program of mobilization and progressive exercise programme for the neck flexors, 2 times a week.
  Arms: Manual Therapy and Exercise
Other: Usual Care (Physiotherapy Intervention) — Active Comparator: Usual Care Participants in this group will receive usual care in physiotherapy during the 6-weeks period.
  Arms: Usual Care

SUMMARY:
The aim of this study is to compare the effectiveness of a combined intervention of manual therapy and exercise versus usual care, on pain intensity, disability, and global perceived recovery, in patients with chronic nonspecific neck pain.

ELIGIBILITY:
Inclusion Criteria:

* Chronic nonspecific neck pain at least 3 months, defined as pain in the cervical region without a specific anatomopathological diagnosis;
* Adults between 18 and 65 years of age and literate in Portuguese;

Exclusion Criteria:

* History of cervical trauma and/or history of surgery in the prior 6 months;
* Clinical signs of infection, tumor, neurological, inflammatory or systemic diseases;
* Pregnancy

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 46 (Estimated)
Dates: Start 2018-06-20 (Estimated); Primary Completion 2018-12 (Estimated); Study Completion 2018-12 (Estimated)

PRIMARY OUTCOMES:
Neck Pain Intensity | Baseline
  Measured using a Numeric Pain Rating Scale (range: 0 - 10 points)
Neck Pain Intensity | 3 weeks
  Measured using a Numeric Pain Rating Scale (range: 0 - 10 points)
Neck Pain Intensity | 6 weeks
  Measured using a Numeric Pain Rating Scale (range: 0 - 10 points)
Neck Pain Intensity | Follow-up 3 months
  Measured using a Numeric Pain Rating Scale (range: 0 - 10 points)
Neck Disability | Baseline
  Measured using the Neck Disability Index (range: 0-50 and higher scores are indicative of more disability)
Neck Disability | 3 weeks
  Measured using the Neck Disability Index (range: 0-50 and higher scores are indicative of more disability)
Neck Disability | 6 weeks
  Measured using the Neck Disability Index (range: 0-50 and higher scores are indicative of more disability)
Neck Disability | Follow-up 3 months
  Measured using the Neck Disability Index (range: 0-50 and higher scores are indicative of more disability)

SECONDARY OUTCOMES:
Neck Global Perceived Recovery | Change from baseline of the global perceived recovery at 3 weeks; 6 weeks; Follow-up 3 months
  Measured using Patient Global Impression of Change Scale to quantify a patient's global improvement over time.

CONTACTS AND LOCATIONS:
Overall Officials: Lúcia Domingues, M.Sc., Principal Investigator — NOVA Medical School | Faculdade de Ciências Médicas, Universidade Nova de Lisboa